CLINICAL TRIAL: NCT05856942
Title: Hybrid Evaluation of the Implementation and Effectiveness of Home-based HIV Pre-exposure Prophylaxis Monitoring in King County, Washington
Brief Title: Hybrid Evaluation of a Home-based HIV Pre-exposure Prophylaxis Program
Acronym: HOT4PrEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Tasso Inc. (Industry)
Responsible Party: Principal Investigator, Chase Cannon, Assistant Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00013871
Record Dates: First submitted 2023-04-06; First posted 2023-05-12 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: HIV Prevention; Pre-exposure Prophylaxis; STI
Keywords: Implementation science; PrEP; Screening; Telehealth
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): Patients will receive standard PrEP care in the clinic including in-person visits for triannual (every 4 months) HIV & STI screening and comprehensive sexual health care.
- Home-based care (Experimental): Patients will have the option to complete their PrEP care from home including 1) self-collection of blood specimens for HIV, syphilis and creatinine; 2) self-swabs for extragenital GC/CT screening; and 3) telehealth follow-up. A maximum of two triannual follow-up visits per year may be conducted remotely; one visit per year must be in person. Participants also have the option to attend visits in person and are otherwise eligible to continue receiving comprehensive sexual health services in the clinic.
  Interventions: Other: Health service - home-based PrEP monitoring

INTERVENTIONS:
Other: Health service - home-based PrEP monitoring — Home-based PrEP care
  Arms: Home-based care

SUMMARY:
The study's aim is to implement a home-based PrEP (HB-PrEP) monitoring system (self-collected blood and extragenital specimens at home and telehealth follow-up) into a large, urban sexual health clinic while also evaluating the program's clinical effectiveness. Study participants will self-collect blood specimens using Tasso devices, which are currently designated as FDA Class 2 exempt medical devices (similar to a medical lancet). This study will be integrated into King County's Ending the HIV Epidemic plan and generate data to inform refinement, adaptation and scale-up of future HB-PrEP programs.

Specific research aims are to:

1. Conduct a hybrid randomized trial to compare the impact of a HB-PrEP program versus standard of care (routine in-clinic monitoring) on PrEP retention over time and use mixed-methods assessments to define the factors that influence HB-PrEP implementation. Hypothesis: HB-PrEP will increase PrEP retention rates by >10% at 18 months and 60% of those offered HB-PrEP will use it for over half of visits.
2. Perform a cost analysis of the HB-PrEP implementation strategy compared to standard care. Hypothesis: HB-PrEP cost will fall within the HIV prevention budget and be affordable with comparable costs to SOC.
3. Develop a qualitative tool to engage healthcare stakeholders and determine the wider scalability of HB-PrEP.

DETAILED DESCRIPTION:
Pre-exposure prophylaxis (PrEP) is an established and effective method for HIV prevention, but lack of access to PrEP providers and the burden of quarterly monitoring visits remain barriers to PrEP uptake and retention, particularly for people of color and younger men who have sex with men (MSM). Home-based PrEP (HB-PrEP) monitoring could unburden medical systems and increase PrEP access, but whether this remote care option improves key clinical outcomes like PrEP retention is not known.

The study's specific aims are to:

* AIM 1: Evaluate the impact of HB-PrEP on PrEP retention and define the factors that influence HB-PrEP implementation. The investigators will conduct a type 1 hybrid randomized controlled trial comparing HB-PrEP as an implementation strategy (self-collected lab specimens from home and telehealth follow-up) to standard of care (SOC) at the Public Health-Seattle & King County (PHSKC) Sexual Health Clinic (SHC). The study's primary outcome will be effectiveness of the implementation strategy measured as the rate of retention in PrEP care. In secondary analyses, investigators will utilize mixed methods to assess reach (proportion of persons offered HB-PrEP who choose to use it), and examine individual-level barriers and facilitators (B&F) to PrEP retention (participant surveys and interviews) and system-level B&F to HB-PrEP implementation (participant surveys and interviews, PHSKC staff interviews). Hypothesis: HB-PrEP will increase PrEP retention rates by >10% at 18 months and 60% of those offered HB-PrEP will use it for over half of visits.
* AIM 2: Perform a cost analysis of HB-PrEP service implementation at the PHSKC SHC compared to SOC. Investigators will track resource use and prospectively collect unit costs for laboratory fees, healthcare worker time and other clinic resources to estimate the total monthly cost of providing HB-PrEP services overall and the monthly cost per person retained in PrEP care in the HB-PrEP and SOC arms. Hypothesis: HB-PrEP cost will fall within the HIV prevention budget and be affordable with comparable costs to SOC.
* AIM 3: Conduct a HB-PrEP scale-up assessment with healthcare organizations (HCO) and other key stakeholders to determine the scalability of HB-PrEP within Washington State. To evaluate institution-level factors that may impede or facilitate statewide HB-PrEP scale-up, investigators will conduct semi-structured interviews with key stakeholders from a countywide EHE HCO collaborative.

The Aim 1 study is a pragmatic, non-blinded, hybrid type 1 (clinical-implementation) RCT and includes mixed-methods assessments to evaluate both qualitative and quantitative data for the primary and secondary outcomes. Aim 3 is a qualitative study using in-depth interviews.

ELIGIBILITY:
Inclusion Criteria:

* Must be eligible to receive PrEP per PHSKC criteria
* Age ≥18 years
* Washington State resident
* Ability to speak, understand and read/write in English or Spanish
* Willing to provide contact information
* Willing to be randomized and adhere to study procedures

Exclusion Criteria:

* Recent (<4 weeks) "high risk" HIV exposure while off PrEP or symptoms of acute HIV
* No mailing address to receive sampling kits
* No working telephone number
* No smartphone or other device with internet access
* History of a bleeding disorder, or current or recent (≤7 days) use of anticoagulant medications
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 458 (Estimated)
Dates: Start 2022-03-08 (Actual); Primary Completion 2025-03-08 (Estimated); Study Completion 2025-09-08 (Estimated)

PRIMARY OUTCOMES:
PrEP retention | 18 months
  Proportion of participants who successfully complete triannual monitoring tests and visits to receive a renewed PrEP prescription

SECONDARY OUTCOMES:
Reach | 18 months
  Proportion of patients who successfully utilize home-based monitoring for at least 50% of triannual visits over the study period
User satisfaction | Every 4 months up to 16 months and at study exit (on/after 18 months)
  Self-reported satisfaction with the assigned PrEP care strategy on Likert scale (1: very satisfied to 5: very dissatisfied)
PrEP adherence | Every 4 months up to 16 months and at study exit (on/after 18 months)
  Self-reported adherence within prior 4 weeks to self-selected PrEP use strategy (daily vs event-driven PrEP); ordinal self-reported adherence scale from excellent to very poor
Time to action on abnormal results | Every 4 months up to 16 months and at study exit (on/after 18 months)
  Time from receipt and review of abnormal monitoring or HIV/STI results to patient notification
STI positivity rate | Every 4 months up to 16 months and at study exit (on/after 18 months)
  Composite asymptomatic STI (syphilis, gonorrhea, chlamydia) rate
Barriers and facilitators of PrEP retention | Every 4 months starting at month 4 until target of 24 reached
  In-depth interviews with study participants and clinic staff/administrators to understand B&F of PrEP retention
Cost | Month 12 through study completion, an average of 6 months
  "Real world" costs of PrEP delivery and retention in each arm (total dollars spent per individual retained on PrEP per month)

CONTACTS AND LOCATIONS:
Overall Officials: Chase Cannon, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Cannon CA, Ramchandani MS, Golden MR. Feasibility of a novel self-collection method for blood samples and its acceptability for future home-based PrEP monitoring. BMC Infect Dis. 2022 May 13;22(1):459. doi: 10.1186/s12879-022-07432-0. PMID 35562692
- [Derived] Cannon C, Holzhauer K, Golden M. Implementation and Evaluation of a Home-Based Pre-Exposure Prophylaxis Monitoring Option: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Sep 23;13:e56587. doi: 10.2196/56587. PMID 39312771